CLINICAL TRIAL: NCT00508742
Title: A Phase 3, Randomized, Active-Controlled, Double-blind Trial Evaluating the Impact of a 13-valent Pneumococcal Conjugate Vaccine on Nasopharyngeal Colonization With Vaccine Serotypes of Streptococcus Pneumoniae in Healthy Infants in Israel.
Brief Title: Study Evaluating the Impact of a 13-valent Pneumococcal Conjugate Vaccine on Nasopharyngeal Colonization
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-3006; B1851007
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2012-07-13 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Pneumococcal Infections
Keywords: Nasopharyngeal Colonization; Streptococcus pneumoniae; Healthy Infants; Vaccines; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 13 valent pneumococcal conjugate vaccine
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- 2 (Active Comparator): 7 valent pneumococcal conjugate vaccine
  Interventions: Biological: 7 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 1 dose at 2, 4, 6 and 12 months of age
  Other Names: 13vPnC
  Arms: 1
Biological: 7 valent pneumococcal conjugate vaccine — 1 dose at 2, 4, 6 and 12 months of age
  Other Names: 7vPnC
  Arms: 2

SUMMARY:
This study is designed to assess the impact of 13-valent Pneumococcal Conjugate Vaccine (13vPnC) on nasopharyngeal colonization with Streptococcus pneumoniae in healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants aged 2 months (42-98 days) at time of enrolment.
* Available for the entire study period and whose parent/legal guardian can be reached by telephone.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with a pneumococcal conjugate vaccine.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1866 (Actual)
Dates: Start 2007-12; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Israel (5):
  - Pfizer Investigational Sites (7), Beersheba, Beer-Sheva
  - Pfizer Investigational Site, Shaqib al-Salam, Segev Shalom
  - Pfizer Investigational Site, Ksaife
  - Pfizer Investigational Site, Rahat
  - Pfizer Investigational Site, Rahat A

REFERENCES:
- [Derived] Dagan R, Jiang Q, Juergens C, Trammel J, Gruber WC, Scott DA. Carrier-Induced Hyporesponsiveness to Pneumococcal Conjugate Vaccines: Unraveling the Influence of Serotypes, Timing, and Previous Vaccine Dose. Clin Infect Dis. 2021 Feb 1;72(3):448-454. doi: 10.1093/cid/ciaa083. PMID 31995183
- [Derived] Dagan R, Juergens C, Trammel J, Patterson S, Greenberg D, Givon-Lavi N, Porat N, Gruber WC, Scott DA. PCV13-vaccinated children still carrying PCV13 additional serotypes show similar carriage density to a control group of PCV7-vaccinated children. Vaccine. 2017 Feb 7;35(6):945-950. doi: 10.1016/j.vaccine.2016.12.052. Epub 2017 Jan 11. PMID 28087146
- [Derived] Dagan R, Juergens C, Trammel J, Patterson S, Greenberg D, Givon-Lavi N, Porat N, Gruber WC, Scott DA. Modeling pneumococcal nasopharyngeal acquisition as a function of anticapsular serum antibody concentrations after pneumococcal conjugate vaccine administration. Vaccine. 2016 Aug 5;34(36):4313-20. doi: 10.1016/j.vaccine.2016.06.075. Epub 2016 Jul 12. PMID 27422342
- [Derived] Dagan R, Juergens C, Trammel J, Patterson S, Greenberg D, Givon-Lavi N, Porat N, Gurtman A, Gruber WC, Scott DA. Efficacy of 13-valent pneumococcal conjugate vaccine (PCV13) versus that of 7-valent PCV (PCV7) against nasopharyngeal colonization of antibiotic-nonsusceptible Streptococcus pneumoniae. J Infect Dis. 2015 Apr 1;211(7):1144-53. doi: 10.1093/infdis/jiu576. Epub 2014 Oct 29. PMID 25355940
- [Derived] Dagan R, Patterson S, Juergens C, Greenberg D, Givon-Lavi N, Porat N, Gurtman A, Gruber WC, Scott DA. Comparative immunogenicity and efficacy of 13-valent and 7-valent pneumococcal conjugate vaccines in reducing nasopharyngeal colonization: a randomized double-blind trial. Clin Infect Dis. 2013 Oct;57(7):952-62. doi: 10.1093/cid/cit428. Epub 2013 Jun 26. PMID 23804191
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3006&StudyName=Study%20Evaluating%20the%20Impact%20of%20a%2013-valent%20Pneumococcal%20Conjugate%20Vaccine%20on%20Nasopharyngeal%20Colonization

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: 13-valent pneumococcal conjugate vaccine (13vPnC) 0.5 milliliter (mL) dose administered intramuscularly at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
- 7vPnC: 7-valent pneumococcal conjugate vaccine (7vPnC) 0.5 mL dose administered intramuscularly at 2, 4, and 6 months of age (infant series) and 12 months of age (toddler dose).
Period: Period 1: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 932 | 934
Vaccinated Dose 1 (at 2 Months of Age) | 930 | 933
Vaccinated Dose 2 (at 4 Months of Age) | 904 | 902
Vaccinated Dose 3 (at 6 Months of Age) | 898 | 892
Completed | 890 | 889
Not Completed | 42 | 45
Not completed — Adverse Event | 5 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Parent/Legal Guardian Request | 31 | 40
Not completed — Physician Decision | 1 | 0
Not completed — Other | 4 | 1
Period: Period 2: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 890 | 889
Completed | 883 | 878
Not Completed | 7 | 11
Not completed — Adverse Event | 2 | 6
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Parent/Legal Guardian Request | 0 | 3
Not completed — Failed to Return | 1 | 0
Not completed — Other | 2 | 1
Period: Period 3: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 883 | 878
Completed | 858 | 863
Not Completed | 25 | 15
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 3
Not completed — Parent/Legal Guardian Request | 17 | 8
Not completed — Other | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 932 | 934 | 1866
Age Continuous [Mean (Standard Deviation); unit: years] | 2.2 (0.3) | 2.2 (0.3) | 2.2 (0.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 474 | 471 | 945
  Male | 458 | 463 | 921

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a New Acquisition of Serotype 6A' (6A + 6C) or 19A Combined 1 Month After the Infant Series to 24 Months of Age
Description: A new acquisition was defined as the detection of a serotype (here 6A' [6A + 6C] or 19A), once a participant was fully vaccinated (one month after dose 3), that had not been detected previously in the baseline samples at 2, 4, 6 months of age.
Time Frame: Month 7 through Month 24
Population: Evaluable culture population included all participants who adhered to protocol requirements; received the treatment to which they were randomized; had at least 1 nasopharyngeal swab for the proposed analysis and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 881 | 873
percentage of participants | 20.0 [17.4 to 22.8] | 36.0 [32.8 to 39.3]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Test type: Superiority or Other; Rate Ratio = 0.56, 95% CI 2-sided [0.47 to 0.65]

2. Secondary Outcome: Percentage of Participants With Nasopharyngeal Cultures Testing Positive for 6A' (6A + 6C) or 19A Serotypes of Streptococcus Pneumoniae (S. Pneumoniae) at 7, 12, 13, 18 and 24 Months of Age
Time Frame: Month 7, 12, 13, 18, 24
Population: Evaluable culture population; 'n' is number of participants with at least 1 determinate nasopharyngeal culture result for given serotype combination at specified time points for each arm group respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 881 | 873
percentage of participants
  Month 7 (n= 881, 871) | 7.3 [5.6 to 9.2] | 10.9 [8.9 to 13.2]
  Month 12 (n= 881, 873) | 8.1 [6.3 to 10.1] | 13.7 [11.5 to 16.2]
  Month 13 (n= 871, 870) | 5.4 [4.0 to 7.1] | 13.6 [11.4 to 16.0]
  Month 18 (n= 864, 864) | 7.1 [5.4 to 9.0] | 13.5 [11.3 to 16.0]
  Month 24 (n= 855, 856) | 6.2 [4.7 to 8.0] | 10.7 [8.8 to 13.0]
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Month 7: 13vPnC/7vPnC, odds ratio was calculated using a logistic regression model with treatment group as the independent variable; Test type: Superiority or Other; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.5 to 0.9]
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Month 12: 13vPnC/7vPnC, odds ratio was calculated using a logistic regression model with treatment group as the independent variable; Test type: Superiority or Other; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.4 to 0.7]
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Month 13: 13vPnC/7vPnC, odds ratio was calculated using a logistic regression model with treatment group as the independent variable; Test type: Superiority or Other; Odds Ratio (OR) = 0.4, 95% CI 2-sided [0.3 to 0.5]
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Month 18: 13vPnC/7vPnC, odds ratio was calculated using a logistic regression model with treatment group as the independent variable; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.4 to 0.7]
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Month 24: 13vPnC/7vPnC, odds ratio was calculated using a logistic regression model with treatment group as the independent variable; Test type: Superiority or Other; Odds Ratio (OR) = 0.5, 95% CI 2-sided [0.4 to 0.8]

ADVERSE EVENTS:
Description: Safety population: all randomized participants with at least 1 dose of study treatment. Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 subject and as nonserious in another, or one subject may have experienced both a serious and nonserious event during study.
Groups:
- Infant Series 13vPnC: Participants who received 13vPnC 0.5 mL intramuscularly at 2, 4 and 6 months of age (infant series), assessed from dose 1 of the infant series through the blood draw 1 month after the infant series.
- Infant Series 7vPnC: Participants who received 7vPnC 0.5 mL intramuscularly at 2, 4 and 6 months of age (infant series), assessed from dose 1 of the infant series through the blood draw 1 month after the infant series.
- After Infant Series 13vPnC: Participants who received 13vPnC 0.5 mL intramuscularly at 2, 4, and 6 months of age in infant series, assessed after the infant series blood draw to the toddler dose.
- After Infant Series 7vPnC: Participants who received 7vPnC 0.5 mL intramuscularly at 2, 4, and 6 months of age in infant series, assessed after the infant series blood draw to the toddler dose.
- Toddler Dose 13vPnC: Participants who received 13vPnC 0.5 mL intramuscularly at 12 months of age (toddler dose), assessed from the toddler dose through the blood draw 1 month after the toddler dose.
- Toddler Dose 7vPnC: Participants who received 7vPnC 0.5 mL dose intramuscularly at 12 months of age (toddler dose), assessed from the toddler dose through the blood draw 1 month after the toddler dose.
- After Toddler Dose 13vPnC: Participants who received 13vPnC 0.5 mL intramuscularly at 12 months of age in toddler dose, assessed after the toddler dose blood draw through the Month 24 visit.
- After Toddler Dose 7vPnC: Participants who received 7vPnC 0.5 mL intramuscularly at 12 months of age in toddler dose, assessed after the toddler dose blood draw through the Month 24 visit.
Arm/Group | Infant Series 13vPnC | Infant Series 7vPnC | After Infant Series 13vPnC | After Infant Series 7vPnC | Toddler Dose 13vPnC | Toddler Dose 7vPnC | After Toddler Dose 13vPnC | After Toddler Dose 7vPnC
Serious Adverse Events (participants affected / at risk) | 64/930 | 57/933 | 48/929 | 64/931 | 15/882 | 23/875 | 91/882 | 73/875
Other Adverse Events (participants affected / at risk) | 454/930 | 433/933 | 290/929 | 324/931 | 238/882 | 240/875 | 462/882 | 455/875
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=930) | Infant Series 7vPnC (N=933) | After Infant Series 13vPnC (N=929) | After Infant Series 7vPnC (N=931) | Toddler Dose 13vPnC (N=882) | Toddler Dose 7vPnC (N=875) | After Toddler Dose 13vPnC (N=882) | After Toddler Dose 7vPnC (N=875)
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cyanosis (Cardiac disorders) | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Ventricular septal defect (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye movement disorder (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Corneal perforation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 2 | 2 | 0 | 1 | 2 | 3
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 2
Oral disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5 | 2 | 0 | 0 | 4 | 14 | 7
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Irritability (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 8 | 4 | 6 | 4 | 0 | 4 | 11 | 10
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Milk allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 10 | 8 | 3 | 4 | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Croup infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysentery (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0 | 4 | 3
Gastroenteritis (Infections and infestations) | 11 | 8 | 12 | 13 | 3 | 4 | 13 | 14
Lower respiratory tract infection (Infections and infestations) | 1 | 4 | 5 | 4 | 0 | 1 | 3 | 1
Meningitis aseptic (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Meningococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 3 | 5 | 9 | 10 | 1 | 3 | 13 | 11
Otitis media acute (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 1 | 3
Pertussis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1 | 5 | 7 | 0 | 1 | 9 | 5
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 3 | 0 | 0 | 3 | 0 | 0 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Rotavirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 1 | 2 | 0 | 2 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 0 | 0 | 0 | 2 | 1
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Exanthema subitum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
Pneumococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Herpangina (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Corynebacterium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endophthalmitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 2 | 1 | 4 | 0 | 2 | 4 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Foreign body (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 2
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza virus test positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 2 | 8 | 6
Diet refusal (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactose intolerance (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeding disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Medulloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 2 | 1 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 2 | 3 | 5 | 1 | 1 | 7 | 8
Fontanelle bulging (Nervous system disorders) | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infantile spasms (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Myoclonic epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cephalhaematoma (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Breath holding (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukocyturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Kidney enlargement (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 3 | 1 | 1 | 2 | 7 | 5
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 0 | 0 | 2
Grunting (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 2 | 1 | 2 | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash macular (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Overfeeding of infant (Social circumstances) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Accidental poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=930) | Infant Series 7vPnC (N=933) | After Infant Series 13vPnC (N=929) | After Infant Series 7vPnC (N=931) | Toddler Dose 13vPnC (N=882) | Toddler Dose 7vPnC (N=875) | After Toddler Dose 13vPnC (N=882) | After Toddler Dose 7vPnC (N=875)
Leukocytosis (Blood and lymphatic system disorders) | 6 | 9 | 13 | 17 | 4 | 4 | 15 | 15
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 2 | 1 | 0 | 2 | 0 | 1 | 1 | 4
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 9 | 13 | 8 | 4 | 7 | 25 | 34
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 2 | 1 | 3 | 13 | 8
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lip swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Swollen tongue (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 4 | 2 | 0 | 0 | 3 | 1 | 0 | 0
Injection site swelling (General disorders) | 14 | 10 | 0 | 0 | 6 | 3 | 0 | 0
Pyrexia (General disorders) | 216 | 194 | 32 | 37 | 90 | 89 | 64 | 68
Developmental delay (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 5 | 3 | 2 | 3 | 0 | 0 | 1 | 5
Bronchiolitis (Infections and infestations) | 1 | 3 | 1 | 1 | 0 | 3 | 5 | 13
Bronchitis (Infections and infestations) | 2 | 5 | 1 | 2 | 1 | 1 | 9 | 10
Cellulitis (Infections and infestations) | 1 | 5 | 1 | 1 | 1 | 2 | 6 | 5
Dysentery (Infections and infestations) | 6 | 4 | 4 | 6 | 1 | 1 | 10 | 13
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 3 | 3 | 2 | 0 | 7 | 3
Infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 2 | 0 | 0 | 1 | 2 | 4
Meningitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 165 | 137 | 176 | 195 | 93 | 92 | 267 | 246
Otitis media acute (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 2
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Investigations) | 12 | 24 | 35 | 32 | 34 | 27 | 112 | 114
Pneumonia (Infections and infestations) | 16 | 14 | 21 | 25 | 7 | 13 | 57 | 58
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 4 | 1 | 0 | 7 | 2
Tonsillitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0 | 2 | 9 | 13
Upper respiratory tract infection (Infections and infestations) | 13 | 5 | 12 | 15 | 2 | 11 | 37 | 43
Urinary tract infection (Infections and infestations) | 11 | 16 | 10 | 5 | 2 | 3 | 10 | 6
Adenoiditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cellulitis orbital (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 6
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pertussis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 3 | 1 | 0 | 0 | 2 | 2
Varicella (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 3
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1
Bullous impetigo (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 5 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Adenoiditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Brucellosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
External ear cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infected bites (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Postoperative fever (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laboratory test (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 3 | 1 | 1 | 0 | 0 | 0 | 0 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight gain poor (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Monarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 5 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Restlessness (Psychiatric disorders) | 98 | 89 | 0 | 0 | 11 | 11 | 1 | 0
Apathy (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 8 | 10 | 4 | 1 | 31 | 20
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 0 | 1 | 3 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 3
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4 | 1 | 0 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Antibiotic prophylaxis (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study designated analysis of effect of 13vPnC on serotypes 6A+19A, changed prior to unblinding, to effect on 6A'+19A. Serotype 6A found to include serotype 6A isolates and isolates of newly identified serotype 6C. Serotype 6A assessed as 6A+6C (6A').

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.